CLINICAL TRIAL: NCT01452217
Title: The Use of Non-invasive MRI to Quantify the Effect of Secretin on Pancreatic Blood Flow and Perfusion in Healthy Volunteers
Brief Title: Non-invasive MRI to Quantify the Effect of Secretin on Pancreatic Blood Flow and Perfusion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D/07/2010
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Pancreatitis
Keywords: Pancreas; Chronic pancreatitis; Perfusion; Blood flow; Magnetic resonance imaging
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secretin (Experimental)
  Interventions: Drug: Secretin

INTERVENTIONS:
Drug: Secretin — Secretin 1 IU/kg over 3 min

SUMMARY:
Alterations in pancreatic blood have been implicated in pancreatic inflammation and pain. Several modalities have been used to assess pancreatic blood flow although some of these methods are invasive, use ionising radiation or intravenous contrast media. This is the first study to utilise non-invasive magnetic resonance imaging to quantify flow within arteries supplying the pancreas and pancreatic perfusion is response to secretin stimulation.

DETAILED DESCRIPTION:
Background An alteration in pancreatic blood flow may be important in a number of clinical conditions. Reduction of blood flow is seen in patients with acute and chronic pancreatitis and the quantification of perfusion may be useful in the management of pancreatic malignancy and assessment of pancreatic transplants. Unfortunately, the measurement of pancreatic blood flow is technically difficult due to the anatomical location of the organ and complex blood supply.

The pancreas receives its blood supply from a rich plexus of arteries but the foremost arterial supply arises from the splenic and pancreaticoduodenal arteries, both superior and inferior.

Various methods have been used in an attempt to quantify the blood flow but all have potential drawbacks. The use of endoscopic and laparoscopic methods are invasive as is the use of intravenous contrast media. Furthermore, the use of computed tomography exposes patients to ionising radiation.

As the arterial supply to the pancreas is complex, measuring single artery flow does not provide an accurate measure of perfusion. Furthermore, as some of the named branches supplying the arteries are secondary or tertiary branches of more major vessels, narrow arterial diameter precludes accurate radiological measurement. Arterial Spin Labelling (ASL) magnetic resonance imaging (MRI), on the other hand is a validated technique allowing accurate measurement of visceral perfusion.

Transient physiological changes occur in pancreatic blood flow secondary to increased demands such as eating. Changes can also be induced pharmacologically using pancreatic stimulating agents, such as secretin. This naturally occuring peptide is produced within the S cells of the proximal small bowel mucosa. It causes an increase in bicarbonate secretion by the duct cells of the pancreas and biliary tract via an oxygen dependant cyclic AMP mediated pathway. Secretin has been used previously to assess alterations in blood flow and is used clinically in the assessment of sphincter of Oddi dysfunction in conjunction with magnetic resonance cholangiopancreatography.

Aims and Hypothesis This pilot study aims to evaluate the MRI techniques of measuring pancreatic perfusion and blood flow at rest and during secretin stimulation in healthy volunteers, prior to an evaluation in the chronic pancreatitis patient group.

Experimental protocol and methods Volunteers will be recruited from advertisements placed on designated University of Nottingham notice boards. All volunteers will complete a questionnaire of abdominal symptoms, Hospital anxiety and depression scale (HAD) and the patient health questionnaire 15 (PhQ15). Each volunteers will attend the 1.5T Brain and Body Imaging centre on the University of Nottingham Campus for all study evaluations.

Following an overnight fast a baseline MRI scan will be undertaken. Volunteers will then receive 1 IU/kg of secretin (Sanochemia Pharmazeutika AG, Wien, Germany) via the intravenous route over 3 minutes.

The volunteers will then be scanned again at 5, 10, 20, 30 and 40 min following the stimulus.

MRI scanning will be carried out on the Philips 1.5T Achieva MRI scanner located in the Brain and Body Imaging Centre University of Nottingham. The volunteers will be placed supine in the scanner with a receiver body coil wrapped around the abdomen. All image analysis will be carried out using commercial and/or in house packages.

Outcome measures at baseline and following secretin stimulation:

1. Pancreatic perfusion
2. Superior mesenteric artery blood flow
3. Gastroduodenal artery blood flow
4. Hepatic artery blood flow
5. Splenic artery blood flow

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Able to give informed consent

Exclusion Criteria:

* Current illness
* Contraindications to magnetic resonance imaging

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pancreatic perfusion | 0, 5, 10, 20, 30 and 40 min
  Overall perfusion of the pancreas

SECONDARY OUTCOMES:
Superior mesenteric artery blood flow | 0, 5, 10, 20, 30 and 40 min
  Blood flow in the superior mesenteric artery
Gastroduodenal artery blood flow | 0, 5, 10, 20, 30 and 40 min
  Blood flow in the gastroduodenal artery
Hepatic artery blood flow | 0, 5, 10, 20, 30 and 40 min
  Blood flow in the hepatic artery
Splenic artery blood flow | 0, 5, 10, 20, 30 and 40 min
  Blood flow in the splenic artery

CONTACTS AND LOCATIONS:
Overall Officials: John Simpson, PhD FRCS, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Delrue L, Blanckaert P, Mertens D, Van Meerbeeck S, Ceelen W, Duyck P. Tissue perfusion in pathologies of the pancreas: assessment using 128-slice computed tomography. Abdom Imaging. 2012 Aug;37(4):595-601. doi: 10.1007/s00261-011-9783-0. PMID 21811851
- [Background] Tsushima Y, Kusano S. Age-dependent decline in parenchymal perfusion in the normal human pancreas: measurement by dynamic computed tomography. Pancreas. 1998 Aug;17(2):148-52. doi: 10.1097/00006676-199808000-00006. PMID 9700945
- [Background] Ishida H, Makino T, Kobayashi M, Tsuneoka K. Laparoscopic measurement of pancreatic blood flow. Endoscopy. 1983 May;15(3):107-10. doi: 10.1055/s-2007-1021480. PMID 6223807
- [Background] Lewis MP, Lo SK, Reber PU, Patel A, Gloor B, Todd KE, Toyama MT, Sherman S, Ashley SW, Reber HA. Endoscopic measurement of pancreatic tissue perfusion in patients with chronic pancreatitis and control patients. Gastrointest Endosc. 2000 Feb;51(2):195-9. doi: 10.1016/s0016-5107(00)70417-2. PMID 10650267
- [Background] Bali MA, Metens T, Denolin V, De Maertelaer V, Deviere J, Matos C. Pancreatic perfusion: noninvasive quantitative assessment with dynamic contrast-enhanced MR imaging without and with secretin stimulation in healthy volunteers--initial results. Radiology. 2008 Apr;247(1):115-21. doi: 10.1148/radiol.2471070685. Epub 2008 Feb 21. PMID 18292476
- [Background] Hacki WH. Secretin. Clin Gastroenterol. 1980 Sep;9(3):609-32. No abstract available. PMID 7000396
- [Background] Bize PE, Platon A, Becker CD, Poletti PA. Perfusion measurement in acute pancreatitis using dynamic perfusion MDCT. AJR Am J Roentgenol. 2006 Jan;186(1):114-8. doi: 10.2214/AJR.04.1416. PMID 16357388
- [Background] Hirota M, Tsuda M, Tsuji Y, Kanno A, Kikuta K, Kume K, Hamada S, Unno J, Ito H, Ariga H, Chiba T, Masamune A, Satoh K, Shimosegawa T. Perfusion computed tomography findings of autoimmune pancreatitis. Pancreas. 2011 Nov;40(8):1295-301. doi: 10.1097/MPA.0b013e31821fcc4f. PMID 21705954
- [Background] Cuthbertson CM, Christophi C. Disturbances of the microcirculation in acute pancreatitis. Br J Surg. 2006 May;93(5):518-30. doi: 10.1002/bjs.5316. PMID 16607683
- [Background] Foitzik T, Eibl G, Hotz HG, Faulhaber J, Kirchengast M, Buhr HJ. Endothelin receptor blockade in severe acute pancreatitis leads to systemic enhancement of microcirculation, stabilization of capillary permeability, and improved survival rates. Surgery. 2000 Sep;128(3):399-407. doi: 10.1067/msy.2000.107104. PMID 10965310
- [Background] Drewes AM, Krarup AL, Detlefsen S, Malmstrom ML, Dimcevski G, Funch-Jensen P. Pain in chronic pancreatitis: the role of neuropathic pain mechanisms. Gut. 2008 Nov;57(11):1616-27. doi: 10.1136/gut.2007.146621. Epub 2008 Jun 19. PMID 18566105
- [Background] Terrace JD, Paterson HM, Garden OJ, Parks RW, Madhavan KK. Results of decompression surgery for pain in chronic pancreatitis. HPB (Oxford). 2007;9(4):308-11. doi: 10.1080/13651820701481497. PMID 18345310
- [Background] Heverhagen JT, Wagner HJ, Ebel H, Levine AL, Klose KJ, Hellinger A. Pancreatic transplants: noninvasive evaluation with secretin-augmented mr pancreatography and MR perfusion measurements--preliminary results. Radiology. 2004 Oct;233(1):273-80. doi: 10.1148/radiol.2331031188. PMID 15454624